CLINICAL TRIAL: NCT02281526
Title: An Open-label, Multiple-dose, Single-centre Study, Investigating the Pharmacokinetics of BIA 2-093 in Subjects With Moderate Hepatic Impairment.
Brief Title: An Open-label, Multiple-dose, Single-centre Study, Investigating the Pharmacokinetics of BIA 2-093
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-111
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with moderate hepatic impairment (Other): This was an open-label, multiple-dose, single-centre study in 2 groups of subjects: subjects with moderate hepatic impairment and healthy controls
  Interventions: Drug: BIA 2-093
- subjects - healthy controls (Other): This was an open-label, multiple-dose, single-centre study in 2 groups of subjects: subjects with moderate hepatic impairment and healthy controls
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: Eslicarbazepine Acetate

SUMMARY:
Open-label, multiple-dose, single-centre study in 2 groups of subjects: subjects with moderate hepatic impairment and healthy controls. The trial consisted of a screening visit, a treatment phase and a follow-up visit. All subjects were to be treated with study medication for 8 consecutive days. Blood and urine were collected for the PK analysis, and safety assessments were performed.

DETAILED DESCRIPTION:
The screening visit was performed 2 to 21 days before the first administration of study medication, the treatment phase consisted of 12 days (of which study medication was administered during the first 8 days), and the follow-up visit was performed 15 to 19 days after the first administration of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age.
* Female subjects had to be post-menopausal, surgically sterilized or using a reliable non-hormonal method of contraception. Examples of reliable non-hormonal methods of contraception include tubal ligation, hysterectomy, intrauterine device, or a barrier method combined with a spermicide. Hormonal contraceptives were not allowed because the effect of BIA 2-093 on the metabolism of oral contraceptives was not yet known.
* Subjects suffering from a chronic illness, other than hepatic impairment, had to have a stable condition, regarded by the investigator as not able to influence the outcome of the study.
* For subjects to be included in Group 1, a stage of moderate hepatic impairment, the extent of which, as measured by the Child-Pugh classification, resulted in recruitment into the study (Group 1 only). This did not apply to subjects that were recruited into Group 2, whose liver functioning was to be normal.
* Body mass not less than 50 kg.

Exclusion Criteria:

* The receipt of any investigational drug within the 30 days prior to this trial.
* Clinically significant abnormal findings (as judged by the investigator) for the following parameters, except those consistent with findings in hepatic impairment: haematology, biochemistry, clotting profile, urinalysis, vital signs or ECG screening tests.
* A history or laboratory evidence of renal impairment and/or disease. Owing to the metabolic pathway of BIA 2-093, any degree of renal impairment would have had a confounding effect on the PK analysis.
* Positive test for Human Immunodeficiency Virus (HIV)-1 or HIV-2 antibodies, Hepatitis B surface antigen and Hepatitis C antibodies. HIV positive patients, and patients with Hepatitis B and C, generally have a below average, and in some cases a markedly decreased, level of health owing to the nature of the respective infections and the natural course of the diseases, both of which are often complicated by an array of opportunistic illnesses. Their ill health would be further worsened by the fact that the patients are hepatically impaired, which has its own, often debilitating, complications. If patients with HIV or Hepatitis B or C were included in the study, this could have led to statistical confusion when assessing the safety and tolerability parameters. This is because events reported by the subjects, which might be a part of the spectrum of complaints in HIV positive patients and Hepatitis B and C patients, would confound the safety and tolerability analysis. In addition, by administering the study medication to these patients, any AEs that might have occurred would add to the discomfort of the patient.
* A history of any illness that, in the opinion of the investigator and/or sponsor, might confound the results of the study or pose additional risk in administering the investigational product to the subject.
* Any planned procedures and/or devices to be performed/added during the course of the study, which might influence the evaluation of the endpoints of the study.
* Current addiction to alcohol as determined by the investigator.
* Use of any medication, prescribed or over-the-counter, except drugs indicated for the treatment of concomitant illnesses in subjects with moderate hepatic impairment, or if the drugs would not have affected the outcome of the study in the opinion of the investigator. Vitamin use was allowed, but should have been stable during the course of the study.
* Current treatment with oxcarbazepine.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Subjects with a supine pulse rate at screening, after resting for 5 min, outside the range of 50 - 100 beats per minute (bpm).
* A history of multiple and/or severe allergies to drugs or foods or a history of anaphylactic reactions.
* Known or suspected allergy to trial product or related products (e.g carbamazepine or oxcarbazepine).
* Female subjects who were pregnant or lactating.
* Previous participation in (recruitment into) this trial.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before dose administration.
* Any history of a bleeding tendency, or an active bleed in the preceding 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Farmovs-Parexel, Bloemfontein, Bloemfontein, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Moderate Hepatic Impairment; Subjects - Healthy Controls: This was an open-label, multiple-dose, single-centre study in 2 groups of subjects: subjects with moderate hepatic impairment and healthy controls
  BIA 2-093
Period: Overall Study
Arm/Group | Subjects With Moderate Hepatic Impairment | Subjects - Healthy Controls
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Moderate Hepatic Impairment | Subjects - Healthy Controls | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve, AUC(0-tlast).
Description: Day 1 - Area under the plasma concentration versus time curve, AUC(0-tlast).
  BIA 2-194, 2-195 Glucoronide, Oxcarbazepine, BIA 2-093 Glucoronide, 2-194 Glucoronide are BIA 2-093 metabolites.
Time Frame: pre-dose and 1, 2, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 7, 9, 12 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: h·ng/mL
Arm/Group | Subjects With Moderate Hepatic Impairment | Subjects - Healthy Controls
Number analyzed (Participants) | 8 | 8
h·ng/mL
  AUC(0-tlast) BIA 2-093 | 954.891 (963.751) | 49.750 (27.931)
  AUC(0-tlast) BIA 2-194 | 240188.369 (27773.762) | 234750.429 (31036.558)
  AUC(0-tlast) 2-195 Glucoronide | 50.603 (44.226) | 157.738 (199.859)
  AUC(0-tlast) Oxcarbazepine | 1489.530 (1055.930) | 1899.092 (915.761)
  AUC(0-tlast) BIA 2-093 Glucoronide | 6.875 (2.312) | 2.500 (2.500)
  AUC(0-tlast) BIA 2-194 Glucoronide | 8634.780 (5915.045) | 11642.372 (11102.059)

2. Secondary Outcome: Cmax - Peak Plasma Concentration
Description: Day 1 - Cmax Peak plasma concentration
Time Frame: pre-dose and 1, 2, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 7, 9, 12 and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Subjects With Moderate Hepatic Impairment | Subjects - Healthy Controls
Number analyzed (Participants) | 8 | 8
ng/mL
  Cmax BIA 2-093 | 477.500 (439.131) | 99.500 (55.861)
  Cmax BIA 2-194 | 16392.778 (3508.757) | 18180.000 (1996.970)
  Cmax 2-195 Glucoronide | 16.875 (19.045) | 16.667 (15.539)
  Cmax Oxcarbazepine | 100.111 (51.948) | 121.000 (63.042)
  Cmax BIA 2-093 Glucoronide | 9.000 (2.449) | 5.000 (5.000)
  Cmax BIA 2-194 Glucoronide | 1067.000 (517.493) | 1381.125 (973.778)

ADVERSE EVENTS:
Arm/Group | Subjects With Moderate Hepatic Impairment | Subjects - Healthy Controls
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/8
Other Adverse Events (participants affected / at risk) | 7/9 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Moderate Hepatic Impairment (N=9) | Subjects - Healthy Controls (N=8)
hepatic encephalopathy (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects With Moderate Hepatic Impairment (N=9) | Subjects - Healthy Controls (N=8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
VOMITING (Gastrointestinal disorders) | 6 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 3
DIZZINESS (Nervous system disorders) | 2 | 0
FATIGUE (General disorders) | 0 | 3
CHILLS (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SCRATCH (Injury, poisoning and procedural complications) | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 2 | 0
BLOOD MAGNESIUM DECREASED (Investigations) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other